CLINICAL TRIAL: NCT05375370
Title: Prediction of Hepatocellular Carcinoma Recurrence After Curative Treatment by Monitoring Circulating Tumor DNA: a Prospective Cohort Study
Brief Title: Prediction of Hepatocellular Carcinoma Recurrence After Curative Treatment by Monitoring Circulating Tumor DNA
Acronym: REMNANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/0414/OB
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: ctDNA; biomarker
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with hepatocellular carcinoma (Experimental): Circulating tumor DNA dosage will be done to patients with hepatocellular carcinoma
  Interventions: Other: circulating tumor DNA dosage

INTERVENTIONS:
Other: circulating tumor DNA dosage — blood sample for circulating tumor DNA dosage will be done to patient with hepatocellular carcinoma

SUMMARY:
The goal of the REMNANT study is to confirm the clinical value of detecting a new biomarker, ctDNA (circulating tumor DNA), in the follow-up of patients with operated liver cancer. In order to meet this objective, this biomarker will be measured in your blood before and after surgery, at three and six months.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer and develops in 80% of cases in the context of underlying cirrhosis1. Surgical resection, percutaneous destruction and liver transplantation are the three treatments considered curative with a non-negligible risk of recurrence of 35-50% at 2 years2.

Several data in the literature suggest that small subclinical tumors can be detected by circulating tumor DNA (ctDNA), and that the amount of tcDNA detected seems to correlate with risk factors for recurrence such as tumor size or microvascular invasion3, 4.

The objective of this pilot study is to evaluate the detection of ctDNA following tumor ablation and its impact on early recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. HCC diagnosed on consensus radiological criteria in cirrhotic patients (EASL-EORTC 2012): helical CT or MRI with triple arterial, portal and late acquisition. The diagnosis is based on the presence of hypervascularization at the early arterial time (wash-in) with wash-out (hypodensity or hypointensity compared to non-tumor liver parenchyma) at the portal phase or late phase compared to non-tumor parenchyma.
3. HCC diagnosed histologically in the absence of a diagnosis on imaging (see IC n°2 above)
4. Patient operated on for liver resection or radiofrequency destruction
5. Treatment decision validated by the digestive oncology PCR
6. Patient having read and understood the information letter and signed the non-opposition form
7. Patient follow-up at the Charles Nicolle University Hospital in Rouen

Exclusion Criteria:

1. Other active cancer or hematological malignancy
2. Contra-indication to surgery
3. Patient not affiliated to the social security system
4. Pregnant woman or parturient or breastfeeding
5. Person under court protection, sub guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change in tcNA dosage between baseline and 6 Months | 6 months
  evolution of tcDNA percentage between Baseline and at 6 months after surgery
Change in tcDNA dosage between baseline and 3 Months | 3 months
  evolution of tcDNA percentage between Baseline and at 3 months after surgery

SECONDARY OUTCOMES:
Survival at 2 years | 2 years
  percentage of Survival 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Edouard ROUSSEL, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Chu Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No